CLINICAL TRIAL: NCT05015101
Title: Evaluation of the Clinical and Radiological Outcome of Uncemented Femoral Stems According to Their Proximal Coating.
Acronym: ETNA
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2019-12-012
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cohort observation — Cohort observation

SUMMARY:
Evaluation of the clinical and radiological outcome of uncemented femoral stems according to their proximal coating.

Retrospective study

DETAILED DESCRIPTION:
On a large population of patients having undergone total hip arthroplasty, divided into two cohorts constituted according to the type of femoral stem implanted (with or without proximal coating by MectaGrip):

Primary objective: To compare between the two groups the radiological osseointegration of the stems five years after arthroplasty.

Secondary objectives: To compare between the groups

* The functional outcome of the arthroplasty
* The frequency of radiological abnormalities (stress shielding, osteolysis, periprosthetic fractures or cracks, periprosthetic ossifications)
* Frequency of complications

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, having been informed of the research
* A patient with at least five years of uncemented total hip replacement implanted as a first-line procedure
* A patient who has been regularly monitored since surgery and for whom all clinical and radiological data are available at the five-year follow-up visit

Exclusion Criteria:

* Patient operated for revision
* History of femoral fracture (pre or per operative)
* Chronic treatment likely to affect calcium metabolism and ossification
* Patient under legal protection, guardianship or curatorship
* A patient who has indicated his or her opposition to the use of his or her medical data (by completing and returning the non-opposition form that will be sent to him or her).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a total hip replacement for at least five years.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-26 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
Engh and Massin Score | 5 years
  The osseointegration of each stem will be assessed by the Engh and Massin score which evaluates the fixation (bone margins and bridges) and the stability of the stem (margins, pedestal, remodelling of the calcar, deterioration of the prosthesis-bone interface, migration, and particles) by associating negative or positive values for each of the parameters. The total constitutes an anatomopathological diagnosis of "confirmed bone rehab" (+ 10 pts and more), suspected (between 0 and + 10 pts), "fibrous encapsulation" (between - 10 and 0 pts) or an "unstable" prosthesis (below - 10 pts).

SECONDARY OUTCOMES:
Stability of the femoral stem: axial migration (sinking) | 5 years
  Radiological assessment of the stability of the femoral stem: axial migration (sinking)
Stability of the femoral stem: frontal migration (varisation) | 5 years
  Radiological assessment of the stability of the femoral stem: frontal migration (varisation)
Gruen's zones assessment | 5 years
  Images of edging, osteolysis, stress shielding according to Gruen's zones
Periprosthetic ossifications (Brooker classification) | 5 years
  Periprosthetic ossifications (Brooker classification)
Periprosthetic fractures (Vancouver classification) | 5 years
  Periprosthetic fractures (Vancouver classification)
Harris Hip Score (HHS) | 5 years
  The Harris Hip Score (HHS) consists of a history part and a clinical examination part that takes into account pain, function and mobility of the hip. A score between 90 and 100 points is defined as excellent, between 80 and 90 as good, between 70 and 80 as fair and below 70 as poor.
Oxford hip score | 5 years
  The Oxford score is a self-assessment of hip joint function consisting of 12 questions scored from 0 to 4. The total score is calculated by adding up the results of each question. The lower the score, the more severe the functional impact.
Forgotten Joint Score | 5 years
  Le Forgotten Joint Score (FJS-12), est un auto-questionnaire compose de 12 questions évaluant le degré d'oubli des prothèses de hanche dans une situation donnée de la vie quotidienne. Chaque réponse est choisie dans une échelle de Likert à 5 points avec les options de réponse allant de jamais (0) la plupart du temps (4).
Life span of prostheses | 5 years
  The life span is the time between the implantation of the prosthesis and its complete or partial surgical revision.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LAUDE, MD PD, Principal Investigator — Clinique du sport
Locations (1):
- Clinique du Sport, Paris, France

IPD SHARING:
Plan to Share IPD: No